CLINICAL TRIAL: NCT04775771
Title: The Effect of Animal-assisted Practice Applied to Hospitalised Children on Children's
Brief Title: The Effect of Animal-assisted Practice Applied to Hospitalised Children on Children's Anxiety, Fear, Psychological and Emotional Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Abdullah Sarman, Lecturer, Inonu University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/1166
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Child Mental Disorder
Keywords: Animal Assisted Practice; Goldfish; Hospitalisation; Anxiety; Fear; Emotional Well-being; Psychological Well-being; Nursing
MeSH Terms: conditions — Neurodevelopmental Disorders; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal Assisted Practice (Experimental) Group (Experimental)
  Interventions: Behavioral: Animal Assisted Practice
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Animal Assisted Practice — The children, who were planned to be hospitalized for at least three days and were randomized to the experimental and control groups, were asked by the researcher using the face-to-face interview technique, and the questions in the patient information form were filled in on the form. Then, pre-test data were recorded by determining their anxiety levels with the State Anxiety Scale for Children, levels of fear with the Child Fear Scale, emotional and psychological well-being with the Stirling Children's Emotional and Psychological Well-being Scale. Unlike the other scales, the anxiety levels were assessed twice with one-hour intervals on the first day with the Children's State Anxiety Scale. On the third day, the anxiety levels were evaluated twice with one-hour intervals on the first day using the State Anxiety Scale for Children. The second group, the children in the control group, had the same procedure except for the intervention; but no intervention was made.
  Arms: Animal Assisted Practice (Experimental) Group

SUMMARY:
In the normal development stage, children become ill for various reasons and maybe hospitalised. Illnesses and hospitalization are major sources of stress for any growing child. In addition to being admitted to the hospital, unknown environment, unknown people in this environment, unknown equipment, scary voices, thought of physical harm, fears such as separation from the family, etc. Different degrees of stress occur for reasons. In addition to these, children face many problems related to physical limitations caused by hospitalization due to illness, and they experience negative emotions such as anxiety, fear, and anxiety. On the day the child is admitted to the hospital, the child and his family experience high levels of anxiety. Children's anxiety and fear may negatively affect their ability to understand the explanations to be made correctly, to interpret events realistically, to make appropriate decisions, and to participate in care. Various treatment methods such as therapeutic games, art therapy, drawing, occupational therapy, animal-assisted practices/activities (HDU) are applied in the hospital environment to improve the child's coping skills and to reduce negative emotions such as pain, anxiety, stress, and fear. The animal-assisted practice is activities that offer various opportunities to improve the quality of life and provide entertainment and therapeutic benefits. Although the use of animal-assisted applications is widespread abroad, its use in our country and the rate of reflection on the results of the study is quite limited. In the researches, interaction with such animals; has been determined to be psychologically, emotionally, socially, and physically supportive in children. It is planned to use goldfish in this study. Aquarium fish is one of the ornamental fish sold in more than 125 countries and more than 2500 species globally. No study has been conducted on the effects of aquarium fish, which are reported to have positive effects and provide calming when applied with adult age groups within the scope of animal-assisted practices, on anxiety, fear, psychological and emotional well-being in children treated in a clinical setting. This study will be conducted to examine the effects of animal-assisted practice on anxiety, fear, the psychological and emotional well-being of children hospitalised.

ELIGIBILITY:
Inclusion Criteria:

* Being 8 years old and over, 10 years old or younger,
* Hospitalization due to an acute illness,
* Not afraid of aquarium fish to be used in practice,
* Not being allergic to fish and fish food,
* Not having physical, auditory, visual, and cognitive disabilities that would prevent the aquarium fish from feeding twice daily and in the aquarium within the scope of HDU,
* Staying in the pediatric clinic for three days,
* Not having a speech disorder that will prevent them from communicating.

Exclusion Criteria:

* Having a physical, auditory, visual, and cognitive disability that prevents the aquarium fish from feeding twice daily,
* Afraid of goldfish,
* Being allergic to fish and eating.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
The mean of STAI-1 | Ten months
  The State Anxiety Inventory for Children (STAI-1): It consists of 20 items scored from 1 to 3 according to the severity and the scores to be obtained from the scale data range between 20 and 60. The Cronbach-Alpha value of the scale was found to be 0.82. Although the validity and reliability study of the scale has been conducted on children aged 9-12, it is also used in children between the ages of 7-17.

SECONDARY OUTCOMES:
The mean of CFS | Ten months
  The Child Fear Scale (CFS): It is a scale consisting of showing five drawn facial expressions ranging from neutral expression (0 points) to "no fear", to a frightened face (4 points) "severe fear". The scale is intended for children aged 5-10 years.

OTHER OUTCOMES:
The mean of SCWBS | Ten months
  Stirling Children's Emotional and Psychological Well-being Scale (SCWBS): It is a scale developed to measure the emotional and psychological well-being levels of children between the ages of 8-15 and is graded between "never" (1 point) and "always" (5 points), consisting of 12 question items, in accordance with the 5-point Likert model. There is no reverse item on the scale. High scores from the scale indicate a high level of emotional and psychological well-being for children. Item-total correlation coefficients of the scale were ranked between 0.57-0.73; the Cronbach-Alpha internal consistency coefficient was calculated as 0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl Obstetrics and Pediatrics Hospital, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No